CLINICAL TRIAL: NCT01695408
Title: Investigating Significant Health Trends in IPF (INSIGHTS-IPF). Nationwide Prospective Registry.
Brief Title: Investigating Significant Health Trends in Idiopathic Pulmonary Fibrosis
Acronym: INSIGHTS-IPF
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: GWT-TUD GmbH (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: INSIGHTS-IPF
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Drug Treatment; Treatment pathways; Clinical routine; Registry; Outcomes; Survival; Patient-related outcomes; Quality of life; Steroids; Azathioprine; N-Acetylcysteine; Pirfenidone; Tyrosine kinase inhibitors; Nintedanib; multicenter; Germany; Safety; Adverse event
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF), a manifestation of chronic progressive fibrosing interstitial pneumonia,ia a rare disease. Current treatment options are limited, and the mean survival time of the newly diagnosed (mostly elderly) patients is only about 2-3 years. As in Europe data are limited on the characteristics and management of such patients, INSIGHTS-IPF was initiated as a new registry that documents newly diagnosed (incident) and prevalent patients with confirmed IPF diagnosis prospectively.The registry will contribute to the optimization of the management of IPF patients in the long term.

DETAILED DESCRIPTION:
INSIGHTS-IPF will report current and comprehensive data on Idiopathic Pulmonary Fibrosis (IPF) in the long-term.

Baseline (cross-sectional part): Description of characteristics of IPF patients in terms of

* key (socio-) demographic data
* IPF risk factors, comorbidities
* methods used for IPF diagnosis
* IPF disease severity and manifestation (including lung function, cardiopulmonary exercise testing and/or exercise capacity if available, laboratory values, biomarkers)
* IPF treatment (detailed information on prescribed drugs and doses; non-pharmacological treatment; listing and score for lung transplantation)
* assessment of patient-related outcomes (PRO) such as quality of life

Follow-up (prospectively up to at least 2 years after inclusion):

* Clinical course of IPF (e.g. in terms of symptoms, lung function, exercise capacity if available)
* Documentation of treatment pathways (switch/add-on/discontinuation of medication), and of non-pharmacological treatment (e.g. start of long term oxygen therapy; new listing for lung transplantation)Outcomes/events (such as acute respiratory worsening, exacerbations, hospitalisation due to any cause and due to IPF, other complications, survival)
* Patient-related outcomes such as quality of life, assessed once a year(for comparison with baseline)
* Resource use for pharmacoeconomic analyses.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent for participation in the registry
* Newly diagnosed (incident) or known (prevalent) IPF (based on diagnosis of treating physician)

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Idiopathic Pulmonary Fibrosis (confirmed diagnosis according to current ATS/ERS guidelines)
Sampling Method: Probability Sample
Enrollment: 1232 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical course of IPF (in terms of symptoms, lung function, survival) | up to 5 years after inclusion

SECONDARY OUTCOMES:
Characteristics of patients with IPF | up to 5 years after inclusion
Treatment pathways | up to 5 years after inclusion
Functionality and quality of life | up to 5 years after inclusion
  St. Georges Respiratory Questionnaire; University of California Shortness of Breath Questionnaire; EuroQuol 5 dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Behr, MD, PhD, Principal Investigator — Ludwig-Maximilian University (LMU) Munich, Med. Clinic V; David Pittrow, MD, PhD, Study Chair — Institute for Clinical Pharmacology, Medical Faculty, Technical University Dresden
Locations (5):
- Germany (5):
  - Institute for Clinical Pharmacology, Medical Faculty, Technical University, Dresden
  - Klinik für Pneumologie, Medizinische Hochschule Hannover, Hanover
  - Pneumologie und Beatmungsmedizin, Thoraxklinik,Universitätsklinikum, Heidelberg
  - Abteilung für Pneumologie Department Innere Medizin, Neurologie und Dermatologie Universitätsklinikum Leipzig AöR, Leipzig
  - V. Med. Clinic, Ludwig-Maximilians-Unviversity, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behr J, Hoeper MM, Kreuter M, Klotsche J, Wirtz H, Pittrow D. [Characteristics and management of idiopathic pulmonary fibrosis: INSIGHTS-IPF registry]. Dtsch Med Wochenschr. 2012 Dec;137(49):2586-8. doi: 10.1055/s-0032-1327244. Epub 2012 Nov 27. German. PMID 23188642
- [Background] Behr J, Hoeper MM, Kreuter M, Klotsche J, Wirtz H, Pittrow D. Investigating significant health trends in idiopathic pulmonary fibrosis (INSIGHTS-IPF): rationale, aims and design of a nationwide prospective registry. BMJ Open Respir Res. 2014 Jan 3;1(1):e000010. doi: 10.1136/bmjresp-2013-000010. eCollection 2014. PMID 25478169
- [Result] Behr J, Kreuter M, Hoeper MM, Wirtz H, Klotsche J, Koschel D, Andreas S, Claussen M, Grohe C, Wilkens H, Randerath W, Skowasch D, Meyer FJ, Kirschner J, Glaser S, Herth FJ, Welte T, Huber RM, Neurohr C, Schwaiblmair M, Kohlhaufl M, Hoffken G, Held M, Koch A, Bahmer T, Pittrow D. Management of patients with idiopathic pulmonary fibrosis in clinical practice: the INSIGHTS-IPF registry. Eur Respir J. 2015 Jul;46(1):186-96. doi: 10.1183/09031936.00217614. Epub 2015 Apr 2. PMID 25837040
- [Result] Kreuter M, Swigris J, Pittrow D, Geier S, Klotsche J, Prasse A, Wirtz H, Koschel D, Andreas S, Claussen M, Grohe C, Wilkens H, Hagmeyer L, Skowasch D, Meyer JF, Kirschner J, Glaser S, Herth FJF, Welte T, Neurohr C, Schwaiblmair M, Held M, Bahmer T, Frankenberger M, Behr J. Health related quality of life in patients with idiopathic pulmonary fibrosis in clinical practice: insights-IPF registry. Respir Res. 2017 Jul 14;18(1):139. doi: 10.1186/s12931-017-0621-y. PMID 28709421
- [Result] Leuschner G, Klotsche J, Kreuter M, Prasse A, Wirtz H, Pittrow D, Frankenberger M, Behr J, Kneidinger N; INSIGHTS-IPF Registry Group. Idiopathic Pulmonary Fibrosis in Elderly Patients: Analysis of the INSIGHTS-IPF Observational Study. Front Med (Lausanne). 2020 Nov 16;7:601279. doi: 10.3389/fmed.2020.601279. eCollection 2020. PMID 33313046
- [Result] Behr J, Prasse A, Wirtz H, Koschel D, Pittrow D, Held M, Klotsche J, Andreas S, Claussen M, Grohe C, Wilkens H, Hagmeyer L, Skowasch D, Meyer JF, Kirschner J, Glaser S, Kahn N, Welte T, Neurohr C, Schwaiblmair M, Bahmer T, Oqueka T, Frankenberger M, Kreuter M. Survival and course of lung function in the presence or absence of antifibrotic treatment in patients with idiopathic pulmonary fibrosis: long-term results of the INSIGHTS-IPF registry. Eur Respir J. 2020 Aug 13;56(2):1902279. doi: 10.1183/13993003.02279-2019. Print 2020 Aug. PMID 32381492
- [Result] Kreuter M, Swigris J, Pittrow D, Geier S, Klotsche J, Prasse A, Wirtz H, Koschel D, Andreas S, Claussen M, Grohe C, Wilkens H, Hagmeyer L, Skowasch D, Meyer JF, Kirschner J, Glaser S, Kahn N, Welte T, Neurohr C, Schwaiblmair M, Held M, Bahmer T, Oqueka T, Frankenberger M, Behr J. The clinical course of idiopathic pulmonary fibrosis and its association to quality of life over time: longitudinal data from the INSIGHTS-IPF registry. Respir Res. 2019 Mar 15;20(1):59. doi: 10.1186/s12931-019-1020-3. PMID 30876420
- See also: Study website — http://insights-ipf.de